CLINICAL TRIAL: NCT03838471
Title: Correlation Between Symptoms of Central Sensitization and Cognitive Behavioral Factors in People With Chronic Shoulder Pain
Brief Title: Cognitive Behavioral Factors and Central Sensitization in Chronic Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Technological Education Institute of Sterea Ellada (Other)
Collaborators: KAT General Hospital (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Eleni Kapreli, Professor, Technological Education Institute of Sterea Ellada
Other Study IDs: PHYSMSC2
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Shoulder Pain
Keywords: CSI; kinesiophobia; Central Nervous System Sensitization; Catastrophizing; Illness Behavior
MeSH Terms: conditions — Kinesiophobia; Illness Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Central sensitization symptoms: This group will contain persons with a clinically relevant degree of symptoms of CS (CSI score ≥40).
- No Central sensitization symptoms: This group will contain persons with a lower degree of symptoms of CS (CSI score < 40).

SUMMARY:
The objective of this study is to examine the relationship between symptoms of central sensitization (CS) and important cognitive behavioral and psychosocial factors in patients with chronic shoulder pain.

DETAILED DESCRIPTION:
Participants, both male and female, with chronic shoulder pain for at least 3 months will be included in the study. They will complete several questionnaires and a functional test. Spearman's correlation will be used to analyze associations between symptoms of CS and pain behavior, functioning, pain, pain catastrophizing, kinesiophobia, and illness perceptions.

Additionally, a between-group analysis will be performed to compare patients with and without clinically relevant symptoms of CS.

ELIGIBILITY:
Inclusion Criteria:

(1)chronic unilateral shoulder pain (Chronic pain will be defined as pain lasting for 3 or more months. Also, pain intensity will be at least 3 on a 0-10 numerical pain rating scale on most days of the last 3 months).

Exclusion Criteria:

1. recent shoulder dislocation (1 year prior) and/or systemic diseases such as rheumatoid arthritis, fibromyalgia and/or polymyalgia rheumatic
2. shoulder pain considered to be originated from the cervical region, and other traumas,
3. neurological dysfunction (ie, multiple sclerosis or stroke), osteoporosis, haemophilia and/or cancer
4. shoulder surgery
5. participants with shoulder pain after post fracture
6. Being pregnant or given birth in the preceding year
7. Overconsumption of alcohol or any other recreational drug2
8. Cognitive impairment
9. inability to provide informed consent and/or complete written questionnaires

If participants use medication with a known influence on the central nervous system (eg, anti-epileptic and antidepressant, analgesics, and/or NSAID's), it should be stable in medication intake for at least 1 month prior to his/her participation to be included in this study (Kuppers et al. 2017). Patients are required to continue usual care at least 6 weeks prior to study participation to obtain a steady state.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 64 participants suffering from chronic unilateral shoulder pain will be recruited from an orthopedic clinic and a chronic pain clinic. Chronic pain will be defined as pain lasting for 3 or more months. Pain intensity will be at least 3 on a 0-10 numerical pain rating scale on most days of the last 3 months. Shoulder pain conditions will include non-specific shoulder pain, subacromial pain sydrome, rotator cuff tendinopathy, instabillity without trauma, SLAP lession, adhesive capsulitis, acromioclavicular pathology and/or shoulder osteoarthritis. Diagnosis will be carried out by a clinician and the criteria will be controlled in a short interview.
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Central sensitization inventory (CSI) | 10 min
  The CSI contains a "part A" of 25 statements related to current health symptoms, indicative of central sensitisation (scored on a 5-point Likert scale ranging from 0-4). A mean score of 40 is the cut off value for central sensitization (Neblett et al 2013). The CSI has proven psychometric strength (Mayer et al 2012; Neblett et al. 2018).
Oxford Shoulder Score (OSS) | 10 min
  The Oxford Shoulder Score (OSS) is a 12-item patient-reported outcomespecifically designed and developed for assessing the impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems. Substantial evidence from clinical studies shows that the PRO has high internal consistency and is a valid and reliable measure of patient well-being. The intraclass correlation has been calculated as 0.83 (Ekeberg,2008 ). In this study, • Self-report functional will be assessed with the Oxford Shoulder Score.
Tampa Scale for Kinesiophobia | 10 min
  To measure kinesiophobia, the Tampa Scale for Kinesiophobia was used. Patients have to score 17 opinions on a 4-point Likert scale (1 = highly disagree, 4 = highly agree). Scores ≥37/68 indicate kinesiophobia. This questionnaire has good internal consistency and test-retest reliability.
Hospital Anxiety and Depression Scale (HADS) | 10 min
  Hospital Anxiety and Depression Scale (HADS) is commonly used to determine the levels of anxiety and depression. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression. A number of researchers have explored HADS data to establish the cut-off points for caseness of anxiety or depression. Bjelland et al (2002)[2] through a literature review of a large number of studies identified a cut-off point of 8/21 for anxiety or depression. For anxiety (HADS-A) this gave a specificity of 0.78 and a sensitivity of 0.9. For depression (HADS-D) this gave a specificity of 0.79 and a sensitivity of 0.83.
Pain Catastrophizing Scale | 10 min
  To measure the extent of pain catastrophizing, we will be used the Pain Catastrophizing Scale, which consists of 13 items exploring pain-related cognition, which the patient has to score on a 5-point Likert scale (0 = not at all, 4 = all the time). Scores ≥30/52 reveal a clinically relevant degree of catastrophizing. This questionnaire is found to have good internal consistency and test-retest reliability, as well as proven construct and criterion validity.
Brief Illness Perception Questionnaire | 3 min
  Patients' illness perceptions will be measured based on the Brief Illness Perception Questionnaire. The patient has to rate 8 statements on a 10-point scale (1-10). The higher the score, the greater is the extent to which the patient's illness perceptions are threatening him or her.
Arm Endurance Test | 5 min
  Pain behavior will be assessed using the arm Endurance Test. This test measured the time the patient could hold both arms horizontally out to the side describing small circles. The tester continued timing while the fingers remained above a line level with the elbow when the arm was dependent (Hardind et al. 1994).
Numeric Pain Rating Scale | 1 min
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain intensity in adults. The most commonly used is the 11-item NPRS. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").The NPRS is a valid and reliable scale to measure pain intensity. In this study, will rate current pain intensity and mean pain intensity durind the past 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni V Kapreli, MSc, PhD, Study Chair — Technological Educational Institute of Sterea Ellada; Paraskevi Bilika, BSc, Principal Investigator — Technological Educational Institute of Sterea Ellada
Locations (1):
- KAT Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huysmans E, Ickmans K, Van Dyck D, Nijs J, Gidron Y, Roussel N, Polli A, Moens M, Goudman L, De Kooning M. Association Between Symptoms of Central Sensitization and Cognitive Behavioral Factors in People With Chronic Nonspecific Low Back Pain: A Cross-sectional Study. J Manipulative Physiol Ther. 2018 Feb;41(2):92-101. doi: 10.1016/j.jmpt.2017.08.007. Epub 2018 Jan 10. PMID 29329739
- [Background] Cuesta-Vargas AI, Neblett R, Chiarotto A, Kregel J, Nijs J, van Wilgen CP, Pitance L, Knezevic A, Gatchel RJ, Mayer TG, Viti C, Roldan-Jimenez C, Testa M, Caumo W, Jeremic-Knezevic M, Luciano JV. Dimensionality and Reliability of the Central Sensitization Inventory in a Pooled Multicountry Sample. J Pain. 2018 Mar;19(3):317-329. doi: 10.1016/j.jpain.2017.11.006. Epub 2017 Dec 2. PMID 29198933
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Adams LM, Turk DC. Psychosocial factors and central sensitivity syndromes. Curr Rheumatol Rev. 2015;11(2):96-108. doi: 10.2174/1573397111666150619095330. PMID 26088211
- [Background] Neblett R, Cohen H, Choi Y, Hartzell MM, Williams M, Mayer TG, Gatchel RJ. The Central Sensitization Inventory (CSI): establishing clinically significant values for identifying central sensitivity syndromes in an outpatient chronic pain sample. J Pain. 2013 May;14(5):438-45. doi: 10.1016/j.jpain.2012.11.012. Epub 2013 Mar 13. PMID 23490634
- [Background] Coronado RA, George SZ. The Central Sensitization Inventory and Pain Sensitivity Questionnaire: An exploration of construct validity and associations with widespread pain sensitivity among individuals with shoulder pain. Musculoskelet Sci Pract. 2018 Aug;36:61-67. doi: 10.1016/j.msksp.2018.04.009. Epub 2018 May 3. PMID 29751194